CLINICAL TRIAL: NCT00429559
Title: Weekly Administration of Topotecan in Combination With Gemcitabine in Patients With Platinum-resistant Ovarian Cancer
Brief Title: Topotecan in Combination With Gemcitabine in Patients With Platinum-resistant Ovarian Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: A.Kalykaki, Hellenic Oncology Research Group
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/06.14
Record Dates: First submitted 2007-01-30; First posted 2007-01-31 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Ovarian Cancer
Keywords: Cancer;; Ovarian cancer;; Recurrent ovarian cancer platinum-resistant
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms | interventions — Topotecan; Gemcitabine

ARMS (1):
- A (Experimental)
  Interventions: Drug: Hycamptin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Hycamptin — 1.75mg/m2 IV on day 1 every week for 3 weeks in cycles of 4 weeks Number of cycles: until progression
  Other Names: Topotecan
Drug: Gemcitabine — Gemcitabine at starting dose of 700 mg/m 2 with increments of 100 mg/m2 IV on day 1 every week for 3 weeks in cycles of four weeks.
  Number of cycles: until progression
  Other Names: Gemzar

SUMMARY:
Topotecan and gemcitabine are drugs globally registered for recurrent ovarian carcinoma. This trial will determine the maximum tolerated dose and the efficacy of this combination administered weekly in patients with platinum -resistant ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed ovarian adenocarcinoma
* Patients had to have received a front-line, platinum- based chemotherapy regimen
* Patients who progressed or whose best response to their most recent platinum-based therapy was less than a partial response will be classified as having platinum-refractory/resistant ovarian cancer. This category also will include patients with disease progression within six months of completing the most recent platinum-based chemotherapy
* Patients had to have at least one bidimensionally measurable and/or evaluable (unidimensionally measurable) target lesion in a non-irradiated area, or increased Ca 125
* A >= 4 weeks interval between their last chemotherapy regimen and the start of study treatment
* Age > 18 years old
* Performance status (WHO) 0-2
* Life expectancy of at least three months
* Adequate bone marrow function (absolute neutrophil count > 1000/mm^3, platelet count > 100000/mm^3, hemoglobin > 9 gr/mm^3)
* Adequate liver (bilirubin < 1.5 times upper limit of normal and SGOT/SGPT < 2 times upper limit of normal) and renal function (creatinine < 2 mg/dl)
* Informed consent

Exclusion Criteria:

* Pregnant or nursing
* Psychiatric illness or social situation that would preclude study compliance
* Other concurrent uncontrolled illness
* Other invasive malignancy within the past 5 years except nonmelanoma skin cancer

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose and the response rate of gemcitabine plus topotecan. | 1year

SECONDARY OUTCOMES:
Toxicity profile | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Kalikaki, MD, Principal Investigator — University Hospital of Crete, Dep of Medical Oncology
Locations (6):
- Greece (6):
  - University Hospital of Crete, Heraklion, Crete
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - "IASO" General Hospital of Athnes, Dep of Medical Oncology, Athens
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - State General Hospital of Larissa, Dep of Medical Oncology, Larissa
  - "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki